CLINICAL TRIAL: NCT06680505
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Phase Ⅱ Clinical Study to Evaluate the Efficacy and Safety of YZJ-1139 Tablets in the Treatment of Primary Chronic Insomnia Disorder
Brief Title: Safety and Efficacy Study of YZJ-1139 in Primary Chronic Insomnia Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YZJ-1139-2-01
Record Dates: First submitted 2024-11-01; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Insomnia Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- YZJ-1139 10mg (Experimental)
  Interventions: Drug: YZJ-1139 10mg
- YZJ-1139 20mg (Experimental)
  Interventions: Drug: YZJ-1139 20mg
- YZJ-1139 40mg (Experimental)
  Interventions: Drug: YZJ-1139 40mg
- YZJ-1139 60mg (Experimental)
  Interventions: Drug: YZJ-1139 60mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YZJ-1139 10mg — YZJ-1139 10mg tablets
  Arms: YZJ-1139 10mg
Drug: YZJ-1139 20mg — YZJ-1139 20mg tablets
  Arms: YZJ-1139 20mg
Drug: YZJ-1139 40mg — YZJ-1139 40mg tablets
  Arms: YZJ-1139 40mg
Drug: YZJ-1139 60mg — YZJ-1139 60mg tablets
  Arms: YZJ-1139 60mg
Drug: Placebo — Match placebo tablets
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of YZJ-1139 in the short-term treatment of primary chronic insomnia, explore the optimal effective dose, and provide the basis for phase III clinical trials

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 to < 65 years.
2. Meet the clinical diagnostic criteria for primary chronic insomnia disorder as defined in ICSD-3 criteria.
3. PSG results for 2 consecutive nights during the run-in period should meet the following conditions:

1) The mean LPS of 2 nights is ≥ 30 min, with the LPS ≥ 15 min for any night; 2) And/or the mean WASO of 2 nights is ≥ 30 min, with neither night ≥20 min; 3) The mean SE of 2 nights is ≤ 85%, with the SE ≤ 87.5% for both nights. 4. During the study, the patient agreed to follow the daily bedtime between 9 and 12 pm , stayed in bed for 6.5-9 hours every night, and agreed to refrain from taking a nap.

5. Female subjects are confirmed to be non-pregnant at screening; both men of reproductive potential and women of childbearing potential should agree to use medically acceptable and effective contraception throughout the study and within 1 month after the end of the study.

6. Understand the study procedures and contents, voluntarily participate in the clinical study and sign the written Informed Consent Form (ICF), have good compliance during participation in the study, and are willing to attend the visits

Exclusion Criteria:

1. Sleep disorders associated with neurological disorders such as depression, anxiety, sleep disorders due to dementia; depression: Hamilton Depression Scale (HAMD) score ≥ 18 or item 3 (suicidal ideation) score of 3 or more; anxiety: Hamilton Anxiety Scale (HAMA) score ≥ 14; dementia: MMSE scale score ≤ 20 for primary school, ≤ 22 for secondary school (including technical secondary school), and ≤ 23 for college (including junior college).
2. Apnea-hypopnea index [AHI] and/or periodic limb movement index [PLMI] > 10 times/hour detected by PSG monitoring during the run-in period.
3. Patients with severe endocrine diseases, blood diseases, cardiovascular and cerebrovascular diseases, autoimmune diseases, respiratory function impairment and other related diseases.
4. Previous history of nervous system disorders such as epilepsy, schizophrenia, bipolar mental disorder, neurodevelopmental retardation, cognitive disorder, narcolepsy, and restless leg syndrome.
5. Receiving any hypnotics, antidepressants, antipsychotics, anticholinergics, memory-enhancing drugs, antihistamines, CYP3A inducers, CYP3A inhibitors within 2 weeks prior to the start of the lead-in PSG.
6. History of drug taking or addiction, which is known through questioning.
7. Have any lifestyle that interferes with the study process or may interfere with sleep: for example, there will be travels across zones within the next 2 weeks or during the study period, or there will be shift work (night and daytime shift).etc.
8. Special occupants who need to operate machinery during the test period, such as professional drivers, high-altitude operators, etc.
9. Subjects who were treated with any other approved or investigational insomnia medication prior to the study, including other orexin receptor inhibitors, or specific herbal preparations, traditional Chinese medicines, and still needed to continue in the study.
10. AST and ALT > 2 × the upper limit of normal (ULN), or Cr > 1.5 × ULN, or white blood cells < lower limit of normal.
11. Hyperthyroidism or hypothyroidism.
12. History of alcohol abuse (defined as regular daily alcohol consumption exceeding the following criteria: approximately 720 mL of beer, or 240 mL of wine, or 60 mL of liquor).
13. History of drug abuse , or positive urine drug screening (screening and/or baseline) for any indicator.
14. Regular daily consumption of excessive tea and coffee drinks.
15. Patients who have participated in other drug clinical trials within the past 3 months, or participated in other research trials during this trial.
16. Pregnant or lactating women.
17. History of allergy to the investigational product or its components.
18. Have other conditions that make the subject unsuitable for participation in the clinical study in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-08-04 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency (SE) monitored by PSG | Baseline , for all subjects: Day 1 / Day 2,Day 13 / Day 14; for 1/5 subjects: Day 27 / Day 28
  SE is the percentage of the subject 's total sleep time versus the monitored time；Changes from baseline (mean of any consecutive 2 days from Day -7 to Day -1) were evaluated separately for all subjects on Day 1 / Day 2, Day 13 / Day 14 of dosing, and for 1/5 subjects in each group on Day 27 / Day 28 of dosing.

SECONDARY OUTCOMES:
Total sleep time (TST), sleep latency (LPS), sleep wake time (WASO), number of sleep awakenings (NAW) monitored by PSG | Baseline ; for all subjects: Day 1 / Day 2, Day 13 / Day 14; for 1/5 subjects: Day 27 / Day 28
  Changes from baseline (mean of any consecutive 2 days from Day -7 to Da y -1) were evaluated separately for all subjects on Day 1 / Day 2, Day 13 / Day 14 of dosing, and for 1/5 subjects in each group on Day 27 / Day 28 of dosing.
Evaluation of Sleep Structures Recorded by PSG Monitoring | Baseline, for all subjects: Day 1, Day 14; for 1/5 subjects: Day 28
  To evaluate changes from baseline on Day 1 and Day 14 of dosing in all subjects and Day 28 of dosing in 1/5 subjects in each group
Subjective Total Sleep Time (sTST), Subjective Sleep Latency (sTSO) Recorded by Sleep Diary | Baseline, for all subjects: Week 1,Week 2, for 1/5 subjects:Week 4
  The mean value at Week 1 and Week 2 for all subjects and the mean value at Week 4 for 1/5 subjects in each group were evaluated for the changes from the baseline value (mean value during the run-in period)
Total sleep time (TST), sleep latency (SL), sleep awakening time (WASO), number of sleep awakenings (NAW) and sleep efficiency (SE) recorded by body movement recorder | Baseline, for all subjects:Week 1,Week 2, for 1/5 subjects:Week 4
  According to the index values measured by body movement recorder, the mean value at Week 1, mean value at Week 2 and mean value at Week 4 of medication for 1/5 subjects in each group were taken from all subjects to evaluate the change values from the baseline values (mean value during run-in period), respectively
Insomnia Severity Index (ISI) | Baseline, for all subjects: Day 14, for 1/5 subjects:Day 28
  Changes from baseline were evaluated separately for all subjects on Day 14 of dosing and for 1/5 subjects in each group on Day 28 of dosing
Rebound evaluation and proportion of rebound patients | Follow-up Period, 7 days after double-blind treatment.
  All subjects should receive body movement recorder test and sleep diary during the follow-up period, and each indicator will be compared with the baseline period. If the baseline value is reached or worse than the baseline value, it is defined as rebound

CONTACTS AND LOCATIONS:
Locations (33):
- China (33):
  - Beijing HuiLongGuan Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Xuanwu Hospital, Capital Medical University, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - The First Hospital of Jilin University, Changchun
  - Hunan Brain Hospital, Changsha
  - Xiangya Hospital, Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Army Specialty Medical Center, Chongqing
  - Guangdong Provincial People's Hospital, Guangzhou
  - Nanfang Hospital of Southern Medical University (Department of Psychiatry), Guangzhou
  - Nanfang Hospital, Southern Medical University (Sleep Medicine Center), Guangzhou
  - The First Affiliated Hospital of Jinan University, Guangzhou
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - The Affiliated Hospital of Jiujiang University, Jiujiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming
  - The First People's Hospital of Yunnan Province, Kunming
  - Jiangxi Provincial Psychiatric Hospital, Nanchang
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing, Nanjing
  - The First People 's Hospital of Nantong, Nantong
  - Qingdao Municipal Hospital, Qingdao
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou
  - Huashan Hospital Affiliated to Fudan University, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - The First Hospital of Hebei Medical University, Shijiazhuang
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Anding Hospital, Tianjin
  - Wuhan Mental Health Center, Wuhan
  - Tangdu Hospital, Fourth Military Medical University, PLA, Xi'an
  - The Second Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - Henan Provincial People's Hospital, Zhengzhou
  - The Affiliated Hospital of Zunyi Medical College, Zunyi